CLINICAL TRIAL: NCT06753370
Title: Experiences of Children and Young People (CYP) With Cerebral Palsy (CP), Their Parents/Caregivers and Healthcare Professionals in Managing Sleep Disordered Breathing (SDB).
Brief Title: Experiences of Managing Sleep Disordered Breathing in Children With Cerebral Palsy.
Acronym: QualSDB_CP
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC24190
Record Dates: First submitted 2024-12-09; First posted 2024-12-31 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Sleep Disordered Breathing (SDB); Cerebral Palsy (CP); Respiratory Support
Keywords: sleep disordered breathing; cerebral palsy; respiratory support; qualitative research
MeSH Terms: conditions — Sleep Apnea Syndromes; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral palsy (CP) refers to a non-progressive movement disorder, which occurs due to damage to the developing brain around the time of birth. Symptoms of sleep disordered breathing (SDB) include noisy breathing during sleep, increased day-time sleepiness and reduced energy levels. In the long term, SDB might have an effect on the brain and learning, as well as putting strain on the heart.

Children with CP have a higher risk of sleep breathing problems compared to typically-developing children. The negative impact of sleep disturbance in children with CP, on their family members/carers' sleep and mental health cannot be understated. Early recognition and management of SDB is important for children with CP to give these children the best possible sleep quality, and to maximise learning potential.

SDB in children with CP is often under-recognised and under-treated. Treatment of SDB in children with CP might involve wearing a mask that delivers pressurised air to hold open a child's airway and make breathing easier when they are asleep. This is called 'respiratory support' which can be continuous pressure (CPAP) or non-invasive ventilation (NIV) which is pressure support with a back-up breathing rate. There is limited knowledge on the appropriate indications or timing to use them. Though respiratory support in children with CP is proven to help with breathing during sleep, its impact on quality of life, number of hospital admissions or frequency of chest infections is unknown.

This study will analyse the experiences of children with CP being managed for SDB, and the views of their carers/parents, and health professionals involved in their care. By undertaking semi-structured interviews, the investigators aim to explore the impact SDB and it's management has on children

DETAILED DESCRIPTION:
The journey and experience of children with CP being managed for SDB can be unique and varied. Hence a qualitive semi-structed interview will offer the best insight into their journey and learn ways to improve the experiences for other children in the future.

The investigators aim to interview;

* Children with CP aged <16 years old, and able to participate in the interview. No lower age limit is defined, as children with CP can have potential underlying learning disability and chronological lower limit age cut off will not be useful in defining ability to engage with study. Instead, each child will be looked at individually with input from parents/carer to determine ability to engage with study.
* Parents/carers of children with CP. There may be times where only the parent/carer is being interviewed as the child is not able to (or does not wish to) engage with the interview. Where both the child with CP and parent/carer are being interviewed, this will be done concurrently.
* Healthcare professionals involved in the management of children with CP and being (or has been) managed with respiratory support for sleep disordered breathing.

The investigators aim to interview 10 children with CP and/or their parents/carer and 10 health professionals, or till no new themes emerge.

The participants for the interview will be identified by the members of the sleep/LTV team and/or by disseminating the study on charity sites and professional membership groups for suitable individuals to contact the research team to express interest.

Those who have confirmed participation in the study will be invited for a single interview either in person or online. Written consent (on paper copy or online) will be gained before the interview. The interview will be conducted as per the relevant interview schedule for children with CP, parents/carers and health professionals. Relevant additional information about the participant will also be documented in the field notes at time of interview.

ELIGIBILITY:
Inclusion Criteria:

- Children and young people with CP and SDB;

* Children and young people aged less than (but not including) 16 years old
* Formal diagnosis of Cerebral Palsy
* Formal diagnosis of Sleep Disordered Breathing (currently or previously managed with respiratory support)
* Able to understand, communicate (with or without aids) and engage with interview (guided by parents/carer opinion on capacity to engage in interview)

Parents/carers of CYP with CP;

* Parents/carer of CYP with CP and SDB being (or has been) managed with respiratory support

Health care professional;

* Professionals (based in community or hospital setting) involved in the management of SDB in CYP with CP

Exclusion Criteria:

* Children and young people with CP and SDB and their parents/carers;

  * CYP with CP on respiratory support for failure to wean as neonate or for Chronic Lung Disease
  * CYP on respiratory support for other neuromuscular or neurodisability conditions
* Health care professional; Nil

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and young people with cerebral palsy who are (or have been) managed with respiratory support for sleep disordered breathing, their parents/carer and health professionals involved in their care.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Themes describing experiences of assessment and management of sleep disordered breathing in children and young people with CP | From enrolment till end of study at 6 months
  Themes describing the experience of children and young people (CYP) with CP in the assessment and management (with respiratory support) of SDB. Emerging themes will be identified through matrix analysis of semi-structured interview (with a phenomenology methodology).
Themes describing experiences of assessment and management of sleep disordered breathing in family members and carers of children with CP. | From enrollment till end of study at 6 months
  Themes describing the experience of family member/carer in the assessment and management (with respiratory support) of SDB in CYP with CP. Emerging themes will be identified through matrix analysis of semi-structured interview (with a phenomenology methodology).
Themes describing experiences of assessment and management of sleep disordered breathing in healthcare professionals of children with CP. | From enrolment till end of study at 6 months
  Themes describing the experience of healthcare professionals in the assessment and management (with respiratory support) of SDB in CYP with CP. Emerging themes will be identified through matrix analysis of semi-structured interview (with a phenomenology methodology).

SECONDARY OUTCOMES:
Facilitators of establishing respiratory support | From enrollment till end of study at 6 months
  Factors which facilitate initiation and establishing respiratory support for SDB in CYP with CP will be identified through matrix analysis of semi-structured interviews for emerging themes (with a phenomenology methodology).
Barriers to establishing respiratory support | From enrollment till end of study at 6 months
  Factors which act as barriers to setting up and establishing respiratory support for SDB in CYP with CP will be identified through matrix analysis of semi-structured interviews for emerging themes (with a phenomenology methodology).
Accessibility to sleep services | From enrollment till end of study at 6 months
  Strategies to improve accessibility to sleep services for managing SDB in CYP with CP will be identified through matrix analysis of semi-structured interviews for emerging themes (with a phenomenology methodology).

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - NHS Lothian, Edinburgh, Edinbrugh
  - Department of Paediatric Respiratory and Sleep Medicine, Royal Hospital for Children and Young People, Edinburgh, Merseyside

IPD SHARING:
Plan to Share IPD: No